CLINICAL TRIAL: NCT06465446
Title: A Phase III Randomized, Open-label, Multicenter Clinical Study of IMM01 (Timdarpacept) in Combiniation With Tiselizumab Versus Physician's Choice Chemotherapy in PD-(L)1-refractory Classical Hodgkin Lymphoma
Brief Title: A Study of IMM01 Plus Tiselizumab Versus Physician's Choice Chemotherapy in PD(L)1-refractory Classical Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMM01-008
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Classic Hodgkin Lymphoma
MeSH Terms: interventions — tislelizumab; Bendamustine Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IMM01 plus Tiselizuma (Experimental): Participants will receive IMM01 (2.0mg/kg) intravenously each week and tislelizumab (200mg) once every 3 weeks in 3-week treatment cycle, for up to 2 years.
  Interventions: Biological: Tislelizumab; Biological: IMM01
- Physician's Choice Chemotherapy (Active Comparator): Participants will receive physician's choice of either bendamustine or gemcitabie.
  Gemciabine: 90 or 120 mg/m^2 on Day 1 and Day 2, IV, 4-week cycle, for up to 6 cycles.
  Gemcitabine: 1000 mg/m^2 on Day 1 and Day 8, IV, 3-week cycle, for up to 6 cycles.
  Interventions: Drug: Bendamustine; Drug: Gemcitabine

INTERVENTIONS:
Biological: Tislelizumab — IV infusion
  Arms: IMM01 plus Tiselizuma
Biological: IMM01 — 2.0mg/kg, IV infusion
  Other Names: Timdarpacept
  Arms: IMM01 plus Tiselizuma
Drug: Bendamustine — IV infusion
  Arms: Physician's Choice Chemotherapy
Drug: Gemcitabine — IV infusion
  Arms: Physician's Choice Chemotherapy

SUMMARY:
The purpose of this study is to compare efficacy of IMM01 plus Tiselizumab with physician's choice chemotherapy of bendamustine or gemcitabine in participants with PD-(L)1-refractory classical Hodgkin Lymphoma. The study will also assess the safety and tolerability of IMM01 plus Tiselizumab. The primary study hypotheses are that IMM01 plus Tiselizuma is superior to physician's choice chemotherapy with respect to progression-free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* Has histologically confirmed diagnosis of classical Hodgkin lymphoma (cHL).
* PD (L)-1 refractory cHL and exhausted all available treatment options with known clinical benefit.
* Has adequate bone marrow reserves and organ functions.

Exclusion Criteria:

* History of central nervous system (CNS) metastases or active CNS involvement.
* Received prior systemic anticancer therapy within 4 weeks before randomization.
* Received prior ani-CD47 or SIRPa treatment.
* History of human immunodeficiency virus (HIV).
* Has an active autoimmune disease that has required systemic treatment in past 2 years except replacement therapy.
* History of severve allergic reactions to any components of trail durg, humanized antibodies or fusion proteins.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) per Lugano 2014 as Assessed by Independent Review Committee (IRC) | approximately 24 months
  PFS is defined as the time from randomization to the first documented disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall Survival (OS) | approximately 36 months
  OS is defined as the time from randomization to death due to any cause.
Duration of Response (DOR) | approximately 24 months
  DOR is defined as the time from the first documented evidence of complete response or partial response until disease progression or death due to any cause, whichever occurs first.
Number of Participants Who Experienced At Least One Adverse Event (AE) | approximately 18 months
  An AE is any untoward medical occurrence in a clinical study participant temporally associated with the use of study intervention, whether or not considered related to the study intervention.